CLINICAL TRIAL: NCT05991076
Title: Feasibility of Activate Bailando, a Community-based Dance Program, on Balance and Social Connectedness for Latino Older Adults
Brief Title: Feasibility of a Community-based Dance Program for Latino Older Adults
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Wisconsin Institute For Healthy Aging (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-0945; EDUC/KINESIOLOGY (Other: UW Madison)
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Mobility Limitation
Keywords: Hispanic/Latinos; Older Adults
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Activate Bailando Dance Program: The Activate Bailando program is a 6-week dance-focused exercise program that focuses on balance and social connectedness for community-dwelling Spanish-speaking older adults.
  Interventions: Other: Latin Dance

INTERVENTIONS:
Other: Latin Dance — The Activate Bailando class is a dance-focused exercise class that is offered once per week for one hour. The program has been developed by dance educators in the Madison area.

SUMMARY:
The objective of this study is to evaluate the feasibility and preliminary effectiveness of Activate Bailando, a 6-week community-based dance class offered in Spanish to older adults. 20 older adults in the Madison, Wisconsin area who are enrolled in Activate Bailando will complete a pre-and post-program test within 10 days for program start and completion.

DETAILED DESCRIPTION:
The primary aim is to evaluate the feasibility of the Activate Bailando program based on measures of recruitment, retention, attendance, and acceptability.

The secondary aim is to evaluate the preliminary effectiveness of the program on metrics of balance, mobility, social connectedness, and fear of falling.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 55
* Willing and able to participate in the Activate Bailando class
* Willing and able to complete data collection before and after the program

Exclusion Criteria:

* Not Being over the age of 55
* Not willing and able to participate in the Activate Bailando class
* Not willing and able to complete data collection before and after the program

Min Age: 55 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Community-dwelling older adults including Spanish-speaking older adults are enrolled in Activate Bailando, a community-based dance class.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Recruitment rate of participants who enroll in the study | Baseline
  A proportion of participants enrolled in the class and those who participate in the data collection will be reported.
Retention rate of participants who enroll and complete the study | Baseline, posttest (up to 7 weeks)
  A proportion of participants who complete the pre data collection, attend at least half of the classes, and complete the post data collection.
Attendance of Class Participation | Posttest (up to 7 weeks)
  Participants will be asked how many classes they attended at the end of the program.
Acceptability of participation in the class | Posttest (up to 7 weeks)
  Participants will be asked what they enjoyed and what they thought could be improved from the class.

SECONDARY OUTCOMES:
Change in University of California Los Angeles (UCLA) Loneliness Scale | Baseline, Posttest (up to 7 weeks)
  A 3-item survey that measures three dimensions of loneliness: relational connectedness, social connectedness, and self-perceived isolation. The scale has three response categories: hardly ever, some of the time, often. The scores of each question are added to give a range of scores from 3 (least lonely) to 9 (most lonely).
Change in Timed Up and Go Results | Baseline, Posttest (up to 7 weeks)
  A mobility test records the time in seconds that it takes the participant to stand up, walk 10 feet (3 meters), walk back, and sit down again. An older adult who takes greater than or equal to 12 seconds to complete the task is at risk of falling.
Change in the 4-stage balance test | Baseline, Posttest (up to 7 weeks)
  A static balance test for 10 seconds in 4 different positions (stand feed side-by-side, place the instep of the foot so it is touching the big toes of the other foot, tandem stand, stand on one foot). The time the participant is able to balance in each position will be recorded in seconds. An older adult who cannot hold the tandem stand for at least 10 seconds is at increased risk of falling.
Changes in Falls Efficacy Scale (Short Version) | Baseline, Posttest (up to 7 weeks)
  A 7-item survey that measures confidence in one's own ability to complete daily activities without falling on a scale of 1-7 where lower scores indicate more extreme confidence.
Changes in Lubben Social Network Scale (LSNS-6) | Baseline, Posttest (up to 7 weeks)
  A 6-item scale that measures social engagement including family and friends. The total score is calculated by finding the sum of all items. For the LSNS-R, the score ranges between 0 and 60, with a higher score indicating more social engagement. For the LSNS-6, the score ranges between 0 and 30, with a higher score indicating more social engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Columna, PhD, Principal Investigator — UW Madison
Locations (1):
- Catholic Multicultural Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No